CLINICAL TRIAL: NCT01311050
Title: A Phase I-II Trial of Capecitabine (Xeloda), Oxaliplatin and Irinotecan in Combination With Bevacizumab in 1st Line Treatment of Metastatic Colorectal Cancer
Brief Title: A Trial of Capecitabine (Xeloda), Oxaliplatin and Irinotecan in Combination With Bevacizumab in 1st Line Treatment of Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2081-068; RAC# 2081-068
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Irinotecan; Bevacizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine (Xeloda), Oxaliplatin, Irinotecan, Bevacizumab — Capecitabine (Xeloda), Oxaliplatin, Irinotecan, Bevacizumab

SUMMARY:
A Phase I-II Trial of Capecitabine (Xeloda), Oxaliplatin and Irinotecan in Combination with Bevacizumab in 1st Line Treatment of Metastatic Colorectal Cancer

DETAILED DESCRIPTION:
A Phase I-II Trial of Capecitabine (Xeloda), Oxaliplatin and Irinotecan in Combination with Bevacizumab in 1st Line Treatment of Metastatic Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed Metastatic Colorectal Cancer

Exclusion Criteria:

* Patients with diagnosis other than Metastatic Colorectal Cancer

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metastatic Colorectal Cancer
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2009-01

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Elshenawy MA, Badran A, Aljubran A, Alzahrani A, Rauf MS, Eldali A, Bazarbashi S. Survival benefit of surgical resection after first-line triplet chemotherapy and bevacizumab in patients with initially unresectable metastatic colorectal cancer. World J Surg Oncol. 2020 Jul 8;18(1):163. doi: 10.1186/s12957-020-01930-8. PMID 32641137
- [Derived] Bazarbashi S, Aljubran A, Alzahrani A, Mohieldin A, Soudy H, Shoukri M. Phase I/II trial of capecitabine, oxaliplatin, and irinotecan in combination with bevacizumab in first line treatment of metastatic colorectal cancer. Cancer Med. 2015 Oct;4(10):1505-13. doi: 10.1002/cam4.497. Epub 2015 Jul 24. PMID 26207614